CLINICAL TRIAL: NCT05618483
Title: Clinical Efficacy of Xylitol Based Nasal Spray for the Treatment of Mild COVID-19 Infection
Brief Title: Xylitol Based Nasal Spray for COVID-19 Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xlear, Inc (Industry)
Collaborators: Metanoic Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-XYLNS-01
Record Dates: First submitted 2022-11-15; First posted 2022-11-16 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Viral Infection
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Randomization to Nasal Spray or Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized 1:1 to receive the Xylitol Based Nasal Spray or a matching saline base placebo. This is a double blinded study. The Nasal Spray Kits will be randomized and allocated to patients in chronological order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): The participants will receive Xylitol based nasal spray
  Interventions: Device: Nasal Spray
- Control (Placebo Comparator): The participants will receive saline based placebo
  Interventions: Device: Nasal Spray

INTERVENTIONS:
Device: Nasal Spray — The nasal spray is made of xylitol and grapefruit seed extract. The spray is antiviral, but there is no data of its clinical efficacy against Covid-19.
  Other Names: Xlear nasal spray

SUMMARY:
Xlear have developed and patented a xylitol containing nasal spray for the treatment of upper-respiratory tract infections. The nasal spray is comprised of xylitol and GSE (Grapefruit Seed extract) which provides antibacterial properties as well as preventing viral adhesion in the nasal passage. Studies into Xlear's antiviral effects on SARS-CoV-2 are currently ongoing but hypothetically, a Xylitol Based Nasal spray may prove to be a useful and inexpensive treatment for COVID-19 infection.

DETAILED DESCRIPTION:
1. BACKGROUND and RATIONALE

In the wake of the Coronavirus disease 2019 (COVID-19) pandemic, worldwide healthcare has rapidly evolved in response. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel virus responsible for COVID-19, which at the most severe end of the spectrum of disease can require hospitalisation or ICU admission. Preventative measures are currently being taken with numerous vaccination programs across the world. However, there is currently no established treatment for mild COVID-19 infection, i.e., symptomatic infection not requiring hospitalisation, which makes up a significant proportion of cases. Xylitol has shown promising results in combating SARS-CoV-2 in vitro and this study aims to explore whether Xlear's Xylitol based Nasal Spray has an effect in vivo.

1.1 COVID-19 Infection SARS-CoV-2 is a positive-sense, single-strand RNA virus comprised of four structural proteins: Nucleocapsid (N) protein, Membrane (M) protein, Spike (S) protein and Envelope (E) protein. These structural proteins play an important role in receptor binding, transcription, replication and assembly of the virus in host cells (Boopathi et al., 2020). The nasal epithelium acts as the primary site for SARS-CoV-2 binding to angiotensin converting enzyme-2 (ACE2) - the receptor responsible for COVID-19 infection (Zhou et al., 2020). With nasal carriage playing a vital role in transmission, drugs administered intranasally could be a viable therapeutic option (Sungnak et al., 2020).

1.2 Drug: Xylitol Xylitol is a sugar alcohol derived from plants. It is used in the dental profession to prevent plaque build-up and inhibit enamel demineralisation by interfering with the metabolism of Streptococcus mutans, causing cell death and thus preventing dental caries (Janakiram et al., 2017). Xylitol not only demonstrates antimicrobial behaviour but can also modulate immunity and contribute to wound healing (Salli et al., 2019).

1.2.1 Xylitol and Respiratory Tract Infections Xylitol's inhibitory effect on Streptococcus mutans growth has prompted more research into its interactions with other nasopharyngeal pathogens responsible for respiratory tract infections. An in vitro study into alpha-haemolytic Streptococcus pneumoniae and beta-haemolytic Streptococci treated with 1% and 5% xylitol showed statistically significant inhibition of growth over a 24-hour incubation period (Kontiokari et al., 1999).

Another team established xylitol's ability to kill coagulase-negative Staphylococcus. 5% xylitol administered to 21 participants compared to a control group using a saline solution showed a significant decrease in Staphylococcus count from 597 colony forming units (CFU) per swab to 99 CFU per swab (Zabner et al., 2000).

1.2.2 Xylitol and Viruses Xylitol's inhibitory effects on bacteria are well documented but little is known regarding its antiviral properties. Dietary xylitol was used to treat influenza A virus in vivo. Mice given a combination of xylitol and red ginseng had 100% survival rate at 33mg/kg/day of xylitol and 60% survival rate at 3.3mg/kg/day after day 14 of infection versus 0% survival rate on PBS (control), red ginseng and xylitol separately. This suggests a synergistic effect between xylitol and red ginseng (Yin et al., 2014).

A study into xylitol and its interactions with human respiratory syncytial virus (hRSV) was conducted in 2015. Xylitol was tested in vitro on a hRSV suspension and in vivo in mice. The in vitro effect of xylitol showed complete inhibition at concentrations of 3.13mg/ml. Xylitol significantly reduced lung viral titres in mice with 3.3mg/kg/d proving the most effective dose (Xu et al., 2016).

1.3 Grapefruit Seed Extract (GSE) Grapefruit seed extract (GSE) is made from grapefruit seeds. It is used as a natural remedy due to its antioxidant and antimicrobial properties (Reagor et al., 2002; Salehi et al., 2019).

1.3.1 GSE and Viruses GSE was tested on multiple viruses to determine if it had any inhibitory effects. GSE exhibited virucidal activity against avian influenza virus (AIV) and Newcastle disease virus (NDV) but not against infectious bursal disease virus (IBDV) (Komura et al., 2019). These findings may be important as AIV and NDV are enveloped viruses like SARS-CoV-2 whilst IBDV is not (Schoeman et al., 2019). It could be hypothesised that GSE could exhibit similar inhibition on SARS-CoV-2.

1.4 Xlear's Xylitol based Nasal Spray Xlear have developed and patented a xylitol containing nasal spray for the treatment of upper-respiratory tract infections. The nasal spray is comprised of xylitol and GSE which provides antibacterial properties as well as preventing viral adhesion in the nasal passage. Studies into Xlear's antiviral effects on SARS-CoV-2 are currently ongoing but hypothetically, a Xylitol Based Nasal spray may prove to be a useful and inexpensive treatment for COVID-19 infection.

1.4.1 Xlear and Coronavirus Xylitol has been shown to exhibit antiviral properties against SARS-CoV-2 in vitro (Bansal et al., 2021; Ferrer et al., 2020).

USA-WAI/2020 strain was prepared and passaged in Vero 76 cells for testing with Xlear (experiment 2) and its components xylitol and GSE separately (experiment 1). GSE 0.2% reduced SARS-CoV-2 from 3.67 log10 CCID50/0.1 mL to undetectable in experiment 1. Xlear in virucidal assays completely inhibited viral infectively at varying concentrations (90%, 80%, 50%) and reduced viral titre by 2.17 log in 20% concentration indicating a dose-dependent response (Appendix 1) (Ferrer et al., 2020). A subsequent study showed statistically significant reduction in viral titres treated with Xlear nasal spray treatment - 4.2 log10 CCID50/0.1mL to 1.7, a reduction of 2.5 log10 CCID50 (Cannon et al., 2020).

A recent private report by Dr Cagno's team in Lausanne (April 2021) has confirmed the viral killing properties of Xlear in 2021 SARS-CoV-2 strains. Viral stocks were grown in Vero E6 cells belonging to two lineages, B1.1.7 and B1.351. Complete inhibition of viral infectivity was observed in 90%, 60% and 20% concentration Xlear virucidal assays for B1.351. Viral infectivity was similarly completely inhibited in B1.17 at 90% and 60% concentration with a 3.06 log reduction at 20% illustrated in Appendix 2.

A case study was conducted on individuals who had taken Xlear as treatment for COVID-19 infection. Participants were required to spray into each nostril four times per day (140 µL per spray). All individuals showed improvement in symptoms with quicker turnarounds from turning positive to negative via COVID-19 reverse transcriptase polymerase chain reaction (RT-PCR) nasal swabs. Importantly, some individuals had relevant co-morbidities such as current smoking status and obesity. Although it is difficult to attribute symptom improvement and viral load decrease to Xlear's spray, it does provide rationale for a double-blind placebo controlled randomised clinical trial (Go et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and providing signed informed consent and ability to adhere to the requirements and restrictions of this protocol;
* Adult aged ≥18 years old with at least two comorbidities: diabetes (type 1 &2), obesity (BMI >30), hypertension, chronic heart disease, chronic pulmonary disease, chronic liver disease.
* Internet access and capability and willingness to participate in audio or audio/video engagements with medical professionals, receive texts, emails, and phone calls from study staff and have a device and reasonable cellular data or other internet access to submit daily study required information using a smart phone, tablet, laptop, or desktop computer during the study period;
* COVID-19 infection confirmed with a laboratory SARS-CoV-2 RT-PCR nasal swab;
* Specimen collected within the past 48 hours;
* Mild COVID-19 symptoms which may include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, lack of taste or smell without shortness of breath

Exclusion Criteria:

* Not fit to consent and unable to follow the protocol;
* Age <18 years;
* Current tracheostomy or laryngectomy;
* Hypersensitivity to the active substance or to any of the excipients;
* Concomitant respiratory therapy such as oxygen or ventilator support. Positive airway pressure for obstructive sleep apnea is permitted if treatment was established with good compliance at least 3 months before enrolment;
* Need for hospitalisation for any reason;
* Inability to safely self-administer nasal spray
* Any clinical contraindications, as judged by the Qualified Medical Practitioner;
* Clinical signs indicative of moderate, severe or critical COVID severity symptoms (as defined by FDA COVID-19 Guidance Document)
* Mentally or neurologically disabled patients who are considered not fit to consent to their participation in the study;
* Lactating, pregnant or planning to become pregnant during the study period;
* Diagnosed with prior COVID-19 infection (>48 hours from the time the test is reported prior to the time of screening).
* No relevant comorbidity or only one comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-28 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Viral load reduction | Day 0 (baseline), Day 2, 4 6 and 8
  The between-groups difference in log-viral load over the total treatment period

SECONDARY OUTCOMES:
Undetectable viral load | baseline to Day 2, 4, 6 and 8
  Proportion of subjects reaching undetectable viral load
Hospitalization requirement | Baseline through Day 8
  The proportion difference in groups requiring hospitalization
Reduction of clinical symptoms score | Baseline through Day 14
  Measurement of modified Jackson score
Tolerability of Nasal Spray | Baseline through Day 14
  Adverse events and discontinuation of nasal spray use
Safety of Nasal Spray | Baseline through Day 14
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan W Rathore, MBBS, Principal Investigator — University of Health Sciences Lahore; Saqib Mahmood, MBBS PhD, Principal Investigator — University of Health Sciences Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bansal S, Jonsson CB, Taylor SL, Figueroa JM, Dugour AV, Palacios C, Vega JC. Iota-carrageenan and xylitol inhibit SARS-CoV-2 in Vero cell culture. PLoS One. 2021 Nov 19;16(11):e0259943. doi: 10.1371/journal.pone.0259943. eCollection 2021. PMID 34797868
- [Result] Boopathi S, Poma AB, Kolandaivel P. Novel 2019 coronavirus structure, mechanism of action, antiviral drug promises and rule out against its treatment. J Biomol Struct Dyn. 2021 Jun;39(9):3409-3418. doi: 10.1080/07391102.2020.1758788. Epub 2020 Apr 30. PMID 32306836
- [Result] Go CC, Pandav K, Sanchez-Gonzalez MA, Ferrer G. Potential Role of Xylitol Plus Grapefruit Seed Extract Nasal Spray Solution in COVID-19: Case Series. Cureus. 2020 Nov 3;12(11):e11315. doi: 10.7759/cureus.11315. PMID 33173650
- [Result] He X, Lau EHY, Wu P, Deng X, Wang J, Hao X, Lau YC, Wong JY, Guan Y, Tan X, Mo X, Chen Y, Liao B, Chen W, Hu F, Zhang Q, Zhong M, Wu Y, Zhao L, Zhang F, Cowling BJ, Li F, Leung GM. Author Correction: Temporal dynamics in viral shedding and transmissibility of COVID-19. Nat Med. 2020 Sep;26(9):1491-1493. doi: 10.1038/s41591-020-1016-z. PMID 32770170
- [Result] Janakiram C, Deepan Kumar CV, Joseph J. Xylitol in preventing dental caries: A systematic review and meta-analyses. J Nat Sci Biol Med. 2017 Jan-Jun;8(1):16-21. doi: 10.4103/0976-9668.198344. PMID 28250669
- [Result] Komura M, Suzuki M, Sangsriratanakul N, Ito M, Takahashi S, Alam MS, Ono M, Daio C, Shoham D, Takehara K. Inhibitory effect of grapefruit seed extract (GSE) on avian pathogens. J Vet Med Sci. 2019 Mar 30;81(3):466-472. doi: 10.1292/jvms.18-0754. Epub 2019 Feb 4. PMID 30713281
- [Result] Kontiokari T, Uhari M, Koskela M. Effect of xylitol on growth of nasopharyngeal bacteria in vitro. Antimicrob Agents Chemother. 1995 Aug;39(8):1820-3. doi: 10.1128/AAC.39.8.1820. PMID 7486925
- [Result] Salehi B, Fokou PVT, Sharifi-Rad M, Zucca P, Pezzani R, Martins N, Sharifi-Rad J. The Therapeutic Potential of Naringenin: A Review of Clinical Trials. Pharmaceuticals (Basel). 2019 Jan 10;12(1):11. doi: 10.3390/ph12010011. PMID 30634637
- [Result] Salli K, Lehtinen MJ, Tiihonen K, Ouwehand AC. Xylitol's Health Benefits beyond Dental Health: A Comprehensive Review. Nutrients. 2019 Aug 6;11(8):1813. doi: 10.3390/nu11081813. PMID 31390800
- [Result] Schoeman D, Fielding BC. Coronavirus envelope protein: current knowledge. Virol J. 2019 May 27;16(1):69. doi: 10.1186/s12985-019-1182-0. PMID 31133031
- [Result] Tom MR, Mina MJ. To Interpret the SARS-CoV-2 Test, Consider the Cycle Threshold Value. Clin Infect Dis. 2020 Nov 19;71(16):2252-2254. doi: 10.1093/cid/ciaa619. No abstract available. PMID 32435816
- [Result] Tu YP, O'Leary TJ. Testing for Severe Acute Respiratory Syndrome-Coronavirus 2: Challenges in Getting Good Specimens, Choosing the Right Test, and Interpreting the Results. Crit Care Med. 2020 Nov;48(11):1680-1689. doi: 10.1097/CCM.0000000000004594. PMID 32826428
- [Result] Xu ML, Wi GR, Kim HJ, Kim HJ. Ameliorating Effect of Dietary Xylitol on Human Respiratory Syncytial Virus (hRSV) Infection. Biol Pharm Bull. 2016;39(4):540-6. doi: 10.1248/bpb.b15-00773. PMID 27040626
- [Result] Yin SY, Kim HJ, Kim HJ. Protective effect of dietary xylitol on influenza A virus infection. PLoS One. 2014 Jan 2;9(1):e84633. doi: 10.1371/journal.pone.0084633. eCollection 2014. PMID 24392148
- [Result] Zabner J, Seiler MP, Launspach JL, Karp PH, Kearney WR, Look DC, Smith JJ, Welsh MJ. The osmolyte xylitol reduces the salt concentration of airway surface liquid and may enhance bacterial killing. Proc Natl Acad Sci U S A. 2000 Oct 10;97(21):11614-9. doi: 10.1073/pnas.97.21.11614. PMID 11027360
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. Addendum: A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Dec;588(7836):E6. doi: 10.1038/s41586-020-2951-z. No abstract available. PMID 33199918
- [Result] Reagor L, Gusman J, McCoy L, Carino E, Heggers JP. The effectiveness of processed grapefruit-seed extract as an antibacterial agent: I. An in vitro agar assay. J Altern Complement Med. 2002 Jun;8(3):325-32. doi: 10.1089/10755530260128014. PMID 12165190
- [Result] Sungnak W, Huang N, Becavin C, Berg M, Queen R, Litvinukova M, Talavera-Lopez C, Maatz H, Reichart D, Sampaziotis F, Worlock KB, Yoshida M, Barnes JL; HCA Lung Biological Network. SARS-CoV-2 entry factors are highly expressed in nasal epithelial cells together with innate immune genes. Nat Med. 2020 May;26(5):681-687. doi: 10.1038/s41591-020-0868-6. Epub 2020 Apr 23. PMID 32327758
- See also: Cannon, M., Westover, J., Bleher, R., Sanchez-Gonzalez, M. and Ferrer, G. In Vitro Analysis of the Anti-viral Potential of nasal spray constituents against SARS-CoV-2. bioRxiv, 2020. doi/10.1101/2020.12.02.408575 — http://www.biorxiv.org/content/10.1101/2020.12.02.408575v3.abstract
- See also: Ferrer, G., Betancourt, A., Go, C., Vazquez, H., Westover, J., Cagno, V., Tapparel, C. and Sanchez-Gonzalez, M. A Nasal Spray Solution of Grapefruit Seed Extract plus Xylitol Displays Virucidal Activity Against SARS-Cov-2 In Vitro. bioRxiv — http://www.biorxiv.org/content/10.1101/2020.11.23.394114v1.abstract